CLINICAL TRIAL: NCT00821353
Title: Sinus Rhythm Maintenance in Patients With Hypertrophic Cardiomyopathy and Atrial Fibrillation - Randomized Comparison of Antiarrhythmic Therapy vs. Radiofrequency Catheter Ablation (SHAARC)
Brief Title: Antiarrhythmic Therapy Versus Catheter Ablation for Atrial Fibrillation in Hypertrophic Cardiomyopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Pawel Derejko M.D. Ph.D., Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N N402 194635; 1.7/IV/08
Record Dates: First submitted 2009-01-11; First posted 2009-01-13 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Atrial Fibrillation; Hypertrophic Cardiomyopathy
Keywords: Atrial fibrillation; Hypertrophic cardiomyopathy; RF ablation; Antiarrhythmic drugs
MeSH Terms: conditions — Atrial Fibrillation; Cardiomyopathy, Hypertrophic | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RFCA (Active Comparator)
  Interventions: Procedure: RF catheter ablation
- Drug (Active Comparator)
  Interventions: Drug: Antiarrhythmic drugs

INTERVENTIONS:
Procedure: RF catheter ablation — RF catheter ablation
  Arms: RFCA
Drug: Antiarrhythmic drugs — One of AA drugs (preferably Amiodarone) and cardioversion in cases of chronic AF
  Arms: Drug

SUMMARY:
Paroxysmal or chronic atrial fibrillation (AF) develops in about 20- 25% of adult patients with hypertrophic cardiomyopathy (HCM) and represents an important complication in the clinical course of the disease, with adverse long-term consequences on functional status and outcome.

Therefore, aggressive therapeutic strategies are indicated to restore and maintain sinus rhythm (SR) in patients with HCM. Nevertheless, pharmacologic prevention of AF recurrence is challenging because of the limited long-term efficacy and potentially hazardous side effects of available treatment options. Currently radiofrequency catheter ablation (RFCA) of AF is successfully used in clinical practice. However, comparison of the efficacy and safety of these two therapeutic options has not been done up till now in randomized manner in this group of patients.

Thus, the aim of the present study is to compare the efficacy and safety of RFCA vs. antiarrhythmic drug therapy in patients with HCM and AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertrophic cardiomyopathy and paroxysmal or chronic atrial fibrillation

Exclusion Criteria:

* Severe hear failure (NYHA IV)
* Left ventricular ejection fraction <0.30
* Left atrial diameter >65 mm
* Age > 70 years
* Contraindication to anticoagulation with warfarin
* Presence of a mechanical prosthetic valve
* Presence of left atrial thrombus on TEE or CT
* Woman currently pregnant
* Renal failure (GFR < 30 ml/min)
* Hepatic failure
* Untreated hypothyroidism or hyperthyroidism
* LVOT gradient > 50 mmHg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Efficacy: Freedom from atrial fibrillation and atrial flutter (>1 min) on or off antiarrhythmic medications. | 1 year

SECONDARY OUTCOMES:
Changes in total symptomatic and asymptomatic AF burden. | 1 year
Incidence of complications. | 1 year
Changes in left atrial diameter and left ventricular function. | 1 year
Changes in level of Nt-pro-BNP. | 1 year
Changes in symptom severity and quality of life. | 1 year
Changes in exercise capacity assessed by cardiopulmonary exercise testing. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Derejko, MD, PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Lidia Chojnowska, MD, PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Lukasz Szumowski, MD, PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Franciszek Walczak, MD, PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland